CLINICAL TRIAL: NCT03183648
Title: A Follow-up Study to Evaluate the Safety for the Patients With ALLO-ASC-DFU Treatment in Phase 2 Clinical Trial of ALLO-ASC-BI-201
Brief Title: A Follow-up Study to Evaluate the Safety of ALLO-ASC-DFU in ALLO-ASC-BI-201 Clinical Trial
Status: Completed | Type: Observational
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALLO-ASC-BI-202
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: ALLO-ASC-DFU — ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells have anti-inflammatory effect and release growth factors such as vascular endothelial growth factor(VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide a new option in treating a burn.
  This tudy is a follow-up study without intervention.
  Other Names:
  Allogenic adipose-derived mesenchymal stem cells

SUMMARY:
This is an open-label follow up study to evaluate the safety for the subjects with ALLO-ASC-DFU treatment in phase 2 clinical trial (ALLO-ASC-BI-201) for 23 months.

DETAILED DESCRIPTION:
This is an open-label follow up study to evaluate the safety for the subjects with ALLO-ASC-DFU treatment in phase 2 clinical trial (ALLO-ASC-BI-201) for 23 months.

ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells have anti-inflammatory effect and release growth factors such as vascular endothelial growth factor(VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide a new option in treating a burn.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are treated with ALLO-ASC-DFU sheet in phase 2 clinical trial of ALLO-ASC-BI-201.
2. A subject who is willing to follow the protocol and provide informed consent on screening, given that the information with respect to the clinical trial is provided.

Exclusion Criteria:

1. Subjects who are considered not suitable for the study by the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject is enrolled who are treated with ALLO-ASC-DFU sheet in phase 2 clinical trial of ALLO-ASC-BI-201
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 24 months
  Evaluation of AE

SECONDARY OUTCOMES:
Vancouver Burn Scar Scale | Every time of visit for follow up to 24 weeks
  Evaluation of Vancouver Burn Scar Scale

CONTACTS AND LOCATIONS:
Overall Officials: Wook Chun, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym university Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No